CLINICAL TRIAL: NCT05939453
Title: A Randomized, Double-Blind, Controlled Trial of Bright Light Therapy on All-Cause Excessive Daytime Sleepiness in Prader-Willi Syndrome
Brief Title: Impact of Bright Light Therapy on Prader-Willi Syndrome
Acronym: PWS-LT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maimonides Medical Center (Other)
Collaborators: Foundation for Prader-Willi Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Study 2022-08-12-MMC
Record Dates: First submitted 2022-12-12; First posted 2023-07-11 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Prader-Willi Syndrome; Excessive Daytime Sleepiness; Hyperphagia; Body Weight; Mood; Behavior
Keywords: Light Therapy; Aberrant Behavior Checklist; Clinical Global Impression- Improvement; Fitbit; Actigraphy reports; Epworth Sleepiness Scale; Hyperphagia Questionnaire (HQCT); Modified Overt Aggression Scale (MOAS)
MeSH Terms: conditions — Prader-Willi Syndrome; Disorders of Excessive Somnolence; Hyperphagia; Body Weight; Behavior | interventions — Ultraviolet Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham Light (Sham Comparator)
  Interventions: Other: Sham Light
- Light Therapy (Experimental)
  Interventions: Other: Bright Light Therapy

INTERVENTIONS:
Other: Sham Light — Sham treatment will be provided from a light box at a distance of at least 70cm but no greater than 90cm.
  Arms: Sham Light
Other: Bright Light Therapy — Bright Light Therapy will be provided using light box with an artificial full spectrum lamp at a distance of at least 70cm but no greater than 90cm.
  Arms: Light Therapy

SUMMARY:
This is a placebo controlled clinical trial to assess the utility of light therapy as a sufficient treatment for excessive daytime sleepiness in patients with Prader-Willi Syndrome

DETAILED DESCRIPTION:
This is a prospective, placebo controlled, open label clinical trial that examines light therapy as a treatment for excessive daytime sleepiness in patients with Prader-Willi syndrome. Subjects are assessed for changes in mood, behavior, body weight, and hyperphagia during visits. All visits are conducted remotely. There are a total of 8 visits occurring over the course of 8 weeks. After the first visit, all study visits occur on a weekly basis.

Individuals between the ages of 6-18 years old with diagnosis of PWS confirmed by genetic testing will be screened for enrolment by the study team.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PWS confirmed by genetic testing
* Score of 12 or above on the Epworth Sleepiness Scale (ESS).

Exclusion Criteria:

* Subjects with an eye condition that could be negatively affected by bright light such as patients with a history of retinal damage or patients needing photosensitizing medications
* A history of previous treatment with LT
* Patients presenting with active psychosis or mania

Ages: 6 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Clinical Global Impression- Improvement (CGI-I) | 8 Weeks
  A positive clinical response will be determined by a rating of 1 or 2 (Very much/Much improved) on the Clinical Global Impression- Improvement (CGI-I) scale at the end of the blinded trial.

SECONDARY OUTCOMES:
Aberrant Behavior Checklist | 8 Weeks
  Consists of 2 subscales; irritability (15 items) and hyperactivity/noncompliance (16 items).
Self-Injury Trauma scale | 8 Weeks
  Scores of 5 or greater were found to be indicative of borderline personality disorder. Part 1 is ranking based on the number of wounds 1=one would (common in a mild self-injurious behavior but rare in a severe case) 2=two or four wounds (common) and 3=five or more wounds (rare). Injury severity is scored on a subjective basis with labels such as "mild" "moderate" and "severe" accompanied by descriptions of the observed state of the anatomy. Part 3 is the Estimate of Current Risk.
Modified Overt Aggression Scale | 8 Weeks
  Four-part behavior rating scale used to evaluate and document the "frequency and severity" of aggressive episodes.[1] The rating scale is made up of four categories; verbal aggression, aggression against objects, aggression against self, and aggression against others

CONTACTS AND LOCATIONS:
Overall Officials: Deepan Singh, MD, Principal Investigator — Maimonides Medical Center
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States

REFERENCES:
- [Background] Rastad C, Ulfberg J, Lindberg P. Improvement in Fatigue, Sleepiness, and Health-Related Quality of Life with Bright Light Treatment in Persons with Seasonal Affective Disorder and Subsyndromal SAD. Depress Res Treat. 2011;2011:543906. doi: 10.1155/2011/543906. Epub 2011 Jun 13. PMID 21747994
- [Background] Videnovic A, Klerman EB, Wang W, Marconi A, Kuhta T, Zee PC. Timed Light Therapy for Sleep and Daytime Sleepiness Associated With Parkinson Disease: A Randomized Clinical Trial. JAMA Neurol. 2017 Apr 1;74(4):411-418. doi: 10.1001/jamaneurol.2016.5192. PMID 28241159
- [Background] Johns MW. A new method for measuring daytime sleepiness: the Epworth sleepiness scale. Sleep. 1991 Dec;14(6):540-5. doi: 10.1093/sleep/14.6.540. PMID 1798888
- [Background] Lassi G, Priano L, Maggi S, Garcia-Garcia C, Balzani E, El-Assawy N, Pagani M, Tinarelli F, Giardino D, Mauro A, Peters J, Gozzi A, Grugni G, Tucci V. Deletion of the Snord116/SNORD116 Alters Sleep in Mice and Patients with Prader-Willi Syndrome. Sleep. 2016 Mar 1;39(3):637-44. doi: 10.5665/sleep.5542. PMID 26446116
- [Background] Pail G, Huf W, Pjrek E, Winkler D, Willeit M, Praschak-Rieder N, Kasper S. Bright-light therapy in the treatment of mood disorders. Neuropsychobiology. 2011;64(3):152-62. doi: 10.1159/000328950. Epub 2011 Jul 29. PMID 21811085
- [Background] Ito T, Yamadera H, Ito R, Endo S. [Effects of bright light on cognitive disturbances in Alzheimer-type dementia]. Nihon Ika Daigaku Zasshi. 1999 Aug;66(4):229-38. doi: 10.1272/jnms.66.229. Japanese. PMID 10466338
- [Background] Srisurapanont K, Samakarn Y, Kamklong B, Siratrairat P, Bumiputra A, Jaikwang M, Srisurapanont M. Blue-wavelength light therapy for post-traumatic brain injury sleepiness, sleep disturbance, depression, and fatigue: A systematic review and network meta-analysis. PLoS One. 2021 Feb 4;16(2):e0246172. doi: 10.1371/journal.pone.0246172. eCollection 2021. PMID 33539446
- [Background] Adhikari P, Pradhan A, Zele AJ, Feigl B. Supplemental light exposure improves sleep architecture in people with type 2 diabetes. Acta Diabetol. 2021 Sep;58(9):1201-1208. doi: 10.1007/s00592-021-01712-y. Epub 2021 Apr 14. PMID 33851274
- [Background] Sene-Fiorese M, Duarte FO, de Aquino Junior AE, Campos RM, Masquio DC, Tock L, de Oliveira Duarte AC, Damaso AR, Parizotto NA, Bagnato VS. The potential of phototherapy to reduce body fat, insulin resistance and "metabolic inflexibility" related to obesity in women undergoing weight loss treatment. Lasers Surg Med. 2015 Oct;47(8):634-42. doi: 10.1002/lsm.22395. Epub 2015 Jul 29. PMID 26220050
- [Background] Patel VP, Patroneva A, Glaze DG, Davis Ms K, Merikle E, Revana A. Establishing the content validity of the Epworth Sleepiness Scale for Children and Adolescents in Prader-Willi syndrome. J Clin Sleep Med. 2022 Feb 1;18(2):485-496. doi: 10.5664/jcsm.9632. PMID 34437052
- [Background] De Cock VC, Diene G, Molinas C, Masson VD, Kieffer I, Mimoun E, Tiberge M, Tauber M. Efficacy of modafinil on excessive daytime sleepiness in Prader-Willi syndrome. Am J Med Genet A. 2011 Jul;155A(7):1552-7. doi: 10.1002/ajmg.a.34047. Epub 2011 Jun 10. PMID 21671379
- [Background] Pullen LC, Picone M, Tan L, Johnston C, Stark H. Cognitive Improvements in Children with Prader-Willi Syndrome Following Pitolisant Treatment-Patient Reports. J Pediatr Pharmacol Ther. 2019 Mar-Apr;24(2):166-171. doi: 10.5863/1551-6776-24.2.166. PMID 31019411
- [Background] Gillett ES, Perez IA. Disorders of Sleep and Ventilatory Control in Prader-Willi Syndrome. Diseases. 2016 Jul 8;4(3):23. doi: 10.3390/diseases4030023. PMID 28933403
- [Background] Fetveit A, Bjorvatn B. Bright-light treatment reduces actigraphic-measured daytime sleep in nursing home patients with dementia: a pilot study. Am J Geriatr Psychiatry. 2005 May;13(5):420-3. doi: 10.1176/appi.ajgp.13.5.420. PMID 15879592
- [Background] Fisher PM, Madsen MK, Mc Mahon B, Holst KK, Andersen SB, Laursen HR, Hasholt LF, Siebner HR, Knudsen GM. Three-week bright-light intervention has dose-related effects on threat-related corticolimbic reactivity and functional coupling. Biol Psychiatry. 2014 Aug 15;76(4):332-9. doi: 10.1016/j.biopsych.2013.11.031. Epub 2013 Dec 19. PMID 24439303
- [Background] Wirz-Justice A, Bader A, Frisch U, Stieglitz RD, Alder J, Bitzer J, Hosli I, Jazbec S, Benedetti F, Terman M, Wisner KL, Riecher-Rossler A. A randomized, double-blind, placebo-controlled study of light therapy for antepartum depression. J Clin Psychiatry. 2011 Jul;72(7):986-93. doi: 10.4088/JCP.10m06188blu. Epub 2011 Apr 5. PMID 21535997
- [Background] McCune AM, Lundgren JD. Bright light therapy for the treatment of night eating syndrome: A pilot study. Psychiatry Res. 2015 Sep 30;229(1-2):577-9. doi: 10.1016/j.psychres.2015.07.079. Epub 2015 Jul 29. PMID 26239768
- [Background] Figueiro MG. Delayed sleep phase disorder: clinical perspective with a focus on light therapy. Nat Sci Sleep. 2016 Apr 6;8:91-106. doi: 10.2147/NSS.S85849. eCollection 2016. PMID 27110143
- [Background] Soreca I. The role of circadian rhythms in Obstructive Sleep Apnea symptoms and novel targets for treatment. Chronobiol Int. 2021 Sep;38(9):1274-1282. doi: 10.1080/07420528.2021.1929281. Epub 2021 May 24. PMID 34027758
- [Background] Stucky B, Clark I, Azza Y, Karlen W, Achermann P, Kleim B, Landolt HP. Validation of Fitbit Charge 2 Sleep and Heart Rate Estimates Against Polysomnographic Measures in Shift Workers: Naturalistic Study. J Med Internet Res. 2021 Oct 5;23(10):e26476. doi: 10.2196/26476. PMID 34609317